CLINICAL TRIAL: NCT02617498
Title: Spray Diathermy Versus Harmonic Scalpel Technique for Hepatic Parenchymal Transection of Living Donor.
Brief Title: Spray Diathermy Versus Harmonic Scalpel Technique for Hepatic Parenchymal Transection
Acronym: LDLT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hepatic transection
Record Dates: First submitted 2015-11-20; First posted 2015-12-01 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: End Stage Liver Disease
Keywords: living donor liver transplantation
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- harmonic scalpel (Active Comparator): parenchymal liver transection was performed either by harmonic scalpel after demarcation of line of transection by intraoperative US and doppler. The clearly exposed vessels were ligated by 5/0 proline or clipped according to their size.
  Interventions: Device: harmonic scalpel
- spray mode diathermy (Active Comparator): parenchymal liver transection was performed either by spray mode diathermy after demarcation of line of transection by intraoperative US and doppler. The clearly exposed vessels were ligated by 5/0 proline or clipped according to their size.
  Interventions: Device: spray mode diathermy

INTERVENTIONS:
Device: harmonic scalpel — parenchymal liver transection was performed either by harmonic scalpel after demarcation of line of transection by intraoperative US and doppler.
  Other Names: Group A
  Arms: harmonic scalpel
Device: spray mode diathermy — parenchymal liver transection was performed either by spray mode diathermy after demarcation of line of transection by intraoperative US and doppler.
  Other Names: Group B
  Arms: spray mode diathermy

SUMMARY:
Consecutive patients, who were treated for end stage liver cirrhosis by LDLT were included in this a prospective study.Patients enrolled in the study divided into two groups according to the day of surgery. The study population was divided into two groups; group (A) Parenchymal liver transection was performed by harmonic scalpel (HS) and group (B) Parenchymal liver transection was performed by spray diathermy (SD).

DETAILED DESCRIPTION:
Consecutive patients, who were treated for end stage liver cirrhosis by LDLT were included in this a prospective study.Patients enrolled in the study divided into two groups according to the day of surgery. The study population was divided into two groups; group (A) Parenchymal liver transection was performed by harmonic scalpel (HS) and group (B) Parenchymal liver transection was performed by spray diathermy (SD).

Donors and recipient were followed up after hospital discharge with laboratory investigation, abdominal ultrasound, MRCP in selected cases every month for the first month, then every 6 months and then every year postoperatively. Follow up visits included clinical examination, laboratory investigation, doses of immunosuppressive, radiological examination, and doppler US.

The primary outcome was the amount of blood loss during transection. Secondary outcomes were operative time, time of transection, speed of transection/minutes , number of ligation used, degree of postoperative injury which assessed by daily liver function, WBC, C reactive protein, pathological changes at the cut surface, postoperative morbidity (including biliary leakage, collection), cost and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients, who were treated for end stage liver cirrhosis by LDLT

Exclusion Criteria:

-

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
the amount of blood loss | 6 hours during operation
  the amount of blood loss

SECONDARY OUTCOMES:
operative time | minutes during operations
number of ligation used, | hours during operations
extent of necrosis at the cut surface | one week postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El Nakeeb, MD, Study Director — Mansoura University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salah T, Sultan AM, Fathy OM, Elshobary MM, Elghawalby NA, Sultan A, Yassen AM, Elsarraf WM, Elmorshedi M, Elsaadany MF, Shiha UA, Wahab MA. Outcome of right hepatectomy for living liver donors: a single Egyptian center experience. J Gastrointest Surg. 2012 Jun;16(6):1181-8. doi: 10.1007/s11605-012-1851-4. Epub 2012 Feb 28. PMID 22370735
- [Result] Wahab MA, Hamed H, Salah T, Elsarraf W, Elshobary M, Sultan AM, Shehta A, Fathy O, Ezzat H, Yassen A, Elmorshedi M, Elsaadany M, Shiha U. Problem of living liver donation in the absence of deceased liver transplantation program: Mansoura experience. World J Gastroenterol. 2014 Oct 7;20(37):13607-14. doi: 10.3748/wjg.v20.i37.13607. PMID 25309092
- [Result] Sultan AM, Salah T, Elshobary MM, Fathy OM, Elghawalby AN, Yassen AM, Elmorshedy MA, Elsadany MF, Shiha UA, Wahab MA. Biliary complications in living donor right hepatectomy are affected by the method of bile duct division. Liver Transpl. 2014 Nov;20(11):1393-401. doi: 10.1002/lt.23964. PMID 25060964
- [Result] El Moghazy WM, Hedaya MS, Kaido T, Egawa H, Uemoto S, Takada Y. Two different methods for donor hepatic transection: cavitron ultrasonic surgical aspirator with bipolar cautery versus cavitron ultrasonic surgical aspirator with radiofrequency coagulator-A randomized controlled trial. Liver Transpl. 2009 Jan;15(1):102-5. doi: 10.1002/lt.21658. PMID 19109835
- [Result] Takatsuki M, Eguchi S, Yamanouchi K, Tokai H, Hidaka M, Soyama A, Miyazaki K, Hamasaki K, Tajima Y, Kanematsu T. Two-surgeon technique using saline-linked electric cautery and ultrasonic surgical aspirator in living donor hepatectomy: its safety and efficacy. Am J Surg. 2009 Feb;197(2):e25-7. doi: 10.1016/j.amjsurg.2008.01.019. Epub 2008 Jul 17. PMID 18639230
- See also: mansoura university — http://www.mans.edu.eg/